CLINICAL TRIAL: NCT00721058
Title: Pre-operative Contrast Enhanced CT to Improve Delineation of the Tumorbed in Radiotherapy for Breast Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Atrium Medical Center (Other); Maasland Hospital (Other); Maastricht University Medical Center (Other)
Responsible Party: L.J. Boersma M.D., Ph.D, Maastro clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Delineation of tumourbed mamma
Record Dates: First submitted 2008-07-22; First posted 2008-07-23 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: Eligible; Operable; Disease; Conserving; Therapy; Visible mass on mammography; Ultrasound > 0.5 cm; Histologically; Proven
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Other: CT-scan

INTERVENTIONS:
Other: CT-scan — A pre-operative CT-scan will be made

SUMMARY:
Rationale: Whole breast irradiation with 50 Gy after lumpectomy has been shown to reduce the local recurrence rate with a factor 3 to 4. An additional boost of 16 Gy to the tumorbed has been shown to improve the local control rate even further. However, this boost dose appears to reduce not only the local recurrences in the tumorbed, but also elsewhere in the breast, suggesting that the boost may not always be delivered at the correct region. In addition, even with the boost dose of 16 Gy, the local recurrence rate in young patients is still quite high - with the majority of recurrences in the tumorbed. Consequently, further improvement of the local control, especially in young women, is still an important aim to pursue, in order to maintain breast conserving therapy (BCT) as an acceptable treatment option in young women. One way to improve local control may be to increase the dose [Young Boost Trial], but also to improve the definition of the tumorbed, i.e. the target volume for boost irradiation.

Objective: The aim of this study is to investigate the effect of incorporating a contrast-enhanced (CE)-CT-thorax in the target volume delineation process on 1) the coverage of the tumorbed by the 85% isodose, 2) the size of the irradiated boost volumes, and 3) the interobserver variation in target volume delineation.

Study design: A CE-CT scan of the thorax will be made prior to surgery, with the patient in radiation treatment position. After breast conserving surgery, patients will be referred for post-operative radiotherapy according to the standard guidelines. Prior to radiotherapy, a standard CT thorax scan will be made for treatment planning.

The planning target volume (PTV) for the boost will be delineated according to the MAASTRO protocol, by three independent observers (PTV-1A-C), using the planning CT only. Delineation of the boost will be repeated after 3D registration of the pre-operative CT scan with the planning CT-scan (PTV-2A-C). Thereafter, consensus will be obtained for the PTV-1A-C and the PTV-2A-C, resulting in one PTV-1 and one PTV-2 for each patient. Radiation treatment plans (RT-plans) will subsequently be designed for PTV-1 and PTV-2. Coverage of the treatment plans by the 85% isodose for both PTV-1- and PTV-2, and the irradiated volumes (percentage of the volume receiving 95% or more (V95)) will be calculated. Patients will be treated with the treatment plan for PTV-2.

Study population: 60 breast cancer patients, to be treated with BCT, with a mass visible on mammography and/or ultrasound > 0.5 cm, without contraindications for a CE-CT-thorax scan will be included.

Intervention: < 3 weeks prior to lumpectomy a CE-CT-thorax scan will be made of the entire thorax, with the patient in the same position as planned during the post-operative radiotherapy. Intravenous contrast will be given according to the standard thorax protocol of MAASTRO clinic.

Main study parameters/endpoints:

Primary endpoints are:

1. The percentage of the PTV-2 receiving < 85% of the dose, if treated with the RT-plan for PTV-1.
2. Difference in V95 for the RT-plan designed for PTV-1- versus for PTV-2. Other endpoints will be interobserver variation, as measured by 1) percent volume overlap; 2) difference in standard deviation of the average PTV-1 and PTV-2; 3) center of mass assay.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will only be included after written informed consent. The preoperative CE-CT-thorax-scan yields little additional radiation exposure, which will however be negligible compared to the radiation treatment to be given because of the breast cancer. In addition, there is a small risk on an allergic reaction to the intravenous contrast, and on renal complications. Therefore, renal function will be checked prior to giving contrast. A kreatinine clearance < 60 ml/min will be a contra-indication for contrast. The pre-operative CT-scan will be made in MAASTRO clinic, requiring an additional visit to MAASTRO clinic. A possible benefit may be that the pre-operative CE-CT thorax may improve the definition of the target volume, and thereby reduce the risk on a local recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for breast conserving therapy i.e. histologically proven breast cancer
* Operable disease
* Visible mass on mammography or ultrasound > 0.5 c

Exclusion Criteria:

* All contra-indications for breast conserving therapy, i.e. previous radiotherapy of the breast, multicentricity, inoperable disease, or too large tumor in a relatively too small breast, pregnancy.
* Contra-indications for intravenous contrast, i.e. iodine allergy, renal malfunction (kreatinine clearance < 60 ml/min), , previous allergic reaction to i.v. contrast, M. Kahler, use of NSAIDs, Diuretics or Metformine.
* Absence of tumor mass > 0.5 cm on conventional mammography or ultrasound

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The percentage of the PTV-2 receiving < 85% of the dose, if treated with the RT-plan for PTV-1. | 1 year

SECONDARY OUTCOMES:
Difference in V95 for the RT-plan designed for PTV-1- versus for PTV-2 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Boersma, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastro clinic, Maastricht, Limburg, Netherlands